CLINICAL TRIAL: NCT01026766
Title: Effects of Heat and Moisture Exchanger in Combination With Air Forced Warming Blankets or Warming Intravenous Solutions on Intraoperative Hypothermia Prevention in Obese and Non Obese Patients During Intravenous Anesthesia
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Clinical Research Ethic Comittee of Botucatu, Botucatu Medical School, UNESP
Other Study IDs: upeclin/HC/FMB-Unesp-32
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Hypothermia
Keywords: Hypothermia; Obesity; Heat and moisture exchanger; Warming blanket; Warming fluids; Gynecological surgery; Intravenous anesthesia; Obese patients; Non obese patients
MeSH Terms: conditions — Hypothermia; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Non obese/ Warming blankets
- Non obese/ Warming intravenous fluids
- Obese/ Warming intravenous fluids
- Obese/ Warming blankets

SUMMARY:
The aim of the present study was to evaluate if the combination of heat and moisture exchanger with air forced warming blankets or warming intravenous fluids prevents intraoperative hypothermia in obese and non obese women under target controlled infusion-total intravenous anaesthesia (TCI-TIVA) during lower abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* women
* 18-65 years old
* gynecologic
* obesity

Exclusion Criteria:

* fever
* endocrine disease
* hypertension
* vasoactive drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty female obese and non obese patients scheduled to gynecologic surgeries were warmed with warming blankets and warming intravenous fluids in association with heat and moisture exchanger.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano A Fernandes, MD, Principal Investigator — Botucatu Medical School
Locations (1):
- College of Medicine of Botucatu, Botucatu, São Paulo, Brazil